CLINICAL TRIAL: NCT02116803
Title: An Open Label, Multi-center, Extension Study to Evaluate Long-term Safety and Tolerability of Dovitinib in Patients With Solid Tumors, Who Continue to Receive Treatment With Dovitinib (TKI258) in Novartis-sponsored, Single Agent Dovitinib Studies, Which Have Fulfilled the Requirements for the Primary Objective, and Are Benefitting From Continued Dovitinib Treatment as Assessed by the Investigator
Brief Title: An Open Label Multi-center Extension Study to Evaluate Long-term Safety/ Tolerability of Dovitinib in Patients With Solid Tumors Who Continue to Receive Treatment With Dovitinib (TKI258) in Novartis-sponsored Single Agent Dovitinib Studies Which Fulfilled the Requirements for the Primary Objective
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2X01B; 2014-000368-17 (EudraCT Number)
Record Dates: First submitted 2014-04-15; First posted 2014-04-17 (Estimated); Results first posted 2018-02-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-01

CONDITIONS: Solid Tumors
Keywords: solid tumors; TKI258; Dovitinib; fulvestrant; cancers with a mass; bulky tumor; nodule; lump; cancer; solid malignancies
MeSH Terms: conditions — Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- dovitinib (Experimental): Participants were given single agent dovitinib starting with last assigned dose and regimen which patient received in parent study. Additional dose modifications were given at the discretion of the investigator based on guidance provided in the protocol and investigative brochure (IB).
  Interventions: Drug: dovitinib
- dovitinib + fulvestrant (Experimental): Participants were given dovitinib and fulvestrant coadministration starting with last assigned dose and regimen which patient received in parent study. Additional dose modifications were at the discretion of the investigator based on guidance provided in the protocol and IB.
  Interventions: Drug: dovitinib; Drug: fulvestrant

INTERVENTIONS:
Drug: dovitinib — Dovitinib was available in two formulations: capsules of 100 mg strength, and tablets of 100 mg strength and taken orally.
  Other Names: TKI258
Drug: fulvestrant — Fulvestrant is generally available as solution for injection in pre-filled syringes containing 250 mg of fulvestrant in 5 mL solution.
  Arms: dovitinib + fulvestrant

SUMMARY:
The study allowed continued safety follow-up of patients who were on single agent dovitinib or dovitinib in combination with fulvestrant treatment in a Novartis-sponsored study which had met its primary endpoint and were benefiting from the treatment as judged by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* patient was currently enrolled in Novartis sponsored study, which had met its endpoint and was receiving single agent oral dovitinib or dovitinib and fulvestrant coadministration
* patient was currently benefiting from treatment with single agent oral dovitinib or dovitinib and fulvestrant coadministration as determined by the guidelines of the parent protocol and according to the investigator's clinical judgment.
* patient had demonstated compliance
* patient had given written informed consent.

Exclusion Criteria:

* patient had been permanently discontinued from oral dovitinib study treatment, either alone or in combination with fulvestrant, in the parent study
* patient was pregnant or nursing at the time of entry
* women of child-bearing potential and male patients with sexual partners of child-bearing potential unwilling to use highly effective methods of contraception during dosing and for a specified duration after stopping study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05-28 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2016-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (2):
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, The Bronx, New York
- Novartis Investigative Site, Salzburg, Austria
- Novartis Investigative Site, Wilrijk, Belgium
- Novartis Investigative Site, Copenhagen, Denmark
- Italy (2):
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Torino, TO
- Novartis Investigative Site, Osaka, Osaka, Japan
- Novartis Investigative Site, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dovitinib | Dovitinib + Fulvestrant
Started | 10 | 2
Completed | 0 | 0
Not Completed | 10 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Progressive disease | 4 | 0
Not completed — Study terminated by sponsor | 2 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all patients who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dovitinib | Dovitinib + Fulvestrant | Total
Number analyzed (Participants) | 10 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (10.55) | 72.0 (14.14) | 62.3 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events of Grades 3 and 4 Severity
Description: Participants with grades 3 and 4 severity adverse events were assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03, unless otherwise specified. AEs are provided by System Organ Class (SOC). A patient with multiple adverse events within a primary system organ class was counted only once in the total row.
Time Frame: Until the last patient discontinued dovitinib up to 30 months
Population: Safety set: the Safety set included all patients who received at least one dose of study medication. Safety set was identical to Full Analysis Set for this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dovitinib | Dovitinib + Fulvestrant
Number analyzed (Participants) | 10 | 2
Participants
  Any Primary system organ class | 6 | 2
  Blood and lymphatic system disorders | 1 | 0
  Cardiac disorders | 2 | 1
  Ear and Labyrinth disorders | 0 | 0
  Endocrine disorders | 0 | 0
  Eye disorders | 0 | 0
  Gastrointestinal disorders | 1 | 0
  General disorders & administration site conditions | 1 | 0
  Infections and Infestations | 1 | 0
  Injury, poisoning and procedural complications | 0 | 0
  Investigations | 2 | 0
  Metabolism and nutrition Disorders | 1 | 0
  Musculoskeletal and connective tissue disorders | 1 | 0
  Neoplasms benign, malignant & Unspecified | 0 | 1
  Nervous system Disorders | 0 | 0
  Psychiatric disorders | 0 | 0
  Respiratory, thoracic and mediastinal disorders | 1 | 0
  Skin and subcutaneous tissue disorders | 0 | 0
  Vascular disorders | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 2.5 years.
Groups:
- Dovitinib+Fulvestrant: Participants were given single agent dovitinib starting with last assigned dose and regimen which patient received in parent study. Additional dose modifications were given at the discretion of the investigator based on guidance provided in the protocol and investigative brochure (IB).
Arm/Group | Dovitinib | Dovitinib+Fulvestrant
Serious Adverse Events (participants affected / at risk) | 4/10 | 2/2
Other Adverse Events (participants affected / at risk) | 9/10 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dovitinib (N=10) | Dovitinib+Fulvestrant (N=2)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
BRADYCARDIA (Cardiac disorders) | 1 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dovitinib (N=10) | Dovitinib+Fulvestrant (N=2)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 1 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 2 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 1
HYPOTHYROIDISM (Endocrine disorders) | 1 | 0
EYE OEDEMA (Eye disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 3 | 0
DIARRHOEA (Gastrointestinal disorders) | 3 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1
ASTHENIA (General disorders) | 1 | 0
FACE OEDEMA (General disorders) | 1 | 0
FATIGUE (General disorders) | 2 | 1
OEDEMA PERIPHERAL (General disorders) | 2 | 0
PYREXIA (General disorders) | 1 | 0
BRONCHITIS (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 2 | 0
CONTUSION (Injury, poisoning and procedural complications) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 1 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 | 0
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 1 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 0
HEADACHE (Nervous system disorders) | 2 | 0
NEURALGIA (Nervous system disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0
RESTLESSNESS (Psychiatric disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 3 | 0
SEBACEOUS GLAND DISORDER (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 1 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.